CLINICAL TRIAL: NCT01601613
Title: A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Comparison of Recombinant Factor VIIa (NovoSeven®) and Standard Haemostatic Replacement Therapy in Patients With Dengue Haemorrhagic Fever
Brief Title: Activated Recombinant Human Factor VII in Patients With Dengue Haemorrhagic Fever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7-3015
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Dengue Haemorrhagic Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFVIIa (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — 100 mcg/kg body weight administered i.v. (into the vein) followed by standard haemostatic replacement therapy (SHRT) at the Investigator's discretion.
  Arms: rFVIIa
Drug: placebo — 100 mcg/kg body weight administered i.v. (into the vein) followed by standard haemostatic replacement therapy (SHRT) at the Investigator's discretion.
  Arms: placebo

SUMMARY:
This trial is conducted in Asia. The aim of this is to investigate the efficacy and safety of activated recombinant human factor VII (rFVIIa) in achieving haemostasis in patients with Dengue haemorrhagic fever (DHF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of Dengue Haemorrhagic Fever (DHF)
* Patients with a clinical diagnosis of DHF Grades II and III8, requiring standard replacement therapy

Exclusion Criteria:

* Patients with a clinical diagnosis of DHF Grade IV
* Known or suspected allergy to trial product or related products
* Known hypersensitivity to mouse, hamster or bovine protein
* Prior treatment with activated recombinant human factor VII

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2001-07; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with evidence of bleeding as assessed at 2 hours after first trial product administration

SECONDARY OUTCOMES:
Proportion of subjects requiring standard haemostatic replacement therapy during 2 hours after first trial product administration
Proportion of subjects with effective haemostatic efficacy at 2 hours after first trial product administration
Coagulation related variables
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Philippines (3):
  - Novo Nordisk Investigational Site, City of Muntinlupa
  - Novo Nordisk Investigational Site, Manila
  - Novo Nordisk Investigational Site, Quezon City
- Thailand (5):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
  - Novo Nordisk Investigational Site, Khon Kaen
  - Novo Nordisk Investigational Site, Pisanulok
  - Novo Nordisk Investigational Site, Ubonratchathani

REFERENCES:
- [Result] Chuansumrit A, Wangruangsatid S, Lektrakul Y, Chua MN, Zeta Capeding MR, Bech OM; Dengue Study Group. Control of bleeding in children with Dengue hemorrhagic fever using recombinant activated factor VII: a randomized, double-blind, placebo-controlled study. Blood Coagul Fibrinolysis. 2005 Nov;16(8):549-55. doi: 10.1097/01.mbc.0000186837.78432.2f. PMID 16269927
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com